CLINICAL TRIAL: NCT05435027
Title: A Phase 1 SARS-CoV-2 Vaccine Study to Assess the Safety and Tolerability of GRT-R912, GRT-R914, and GRT-R918 Administered as Prime and/or Boost in Healthy Adult Participants and People Living With HIV
Brief Title: Study of Self-Amplifying Messenger Ribonucleic Acid (samRNA) Vaccines Against COVID-19 in Healthy Adults and People Living With Human Immunodeficiency Virus (HIV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gritstone bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GO-012
Record Dates: First submitted 2022-06-24; First posted 2022-06-28 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: SARS-CoV-2 vaccine; Coronavirus Disease (COVID-19); Self-amplifying mRNA (samRNA); Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — COVID-19; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GRT-R914, HIV-negative (Part A) (Experimental): Participants in this ≥18 to 65-year-old Part A are naïve to SARS-CoV-2 (Cohorts A1, A2, and A3) or SARS-CoV-2 convalescent (Cohorts A4, A5, A6). Cohorts will receive doses of GRT-R914 administered as prime and boost on Days 1 and Day 29, or as boost 6 months after primary SARS-CoV-2 infection.
  Interventions: Drug: GRT-R914, samRNA-Spikebeta-TCE9
- GRT-R912, HIV-negative (Part B) (Experimental): Participants in this ≥18 to 65-year-old Part B are naïve to SARS-CoV-2 (Cohorts B1, B2) or SARS-CoV-2 convalescent (Cohorts B3, B4). Cohorts will receive doses of GRT-R912 administered as prime and boost on Days 1 and 29, or as boost 6 months after primary SARS-CoV-2 infection. Parts B, C, and D will be run in parallel.
  Interventions: Drug: GRT-R912, samRNA-Spikebeta-TCE11
- GRT-R912 or GRT-R914, People Living with HIV (PLWH) (Part C) (Experimental): Participants in this ≥18 to 65-year-old Part C are people living with HIV but naïve to SARS-CoV-2 (Cohorts C1, C4) or living with HIV but SARS-CoV-2 convalescent (Cohorts C2, C3, C5, C6). Cohorts will receive doses of GRT-R912 or GRT-R914 administered as prime and boost on Days 1 and 29, or as boost 6 months after primary SARS-CoV-2 infection. Parts B, C, and D will be run in parallel.
  Interventions: Drug: GRT-R912, samRNA-Spikebeta-TCE11; Drug: GRT-R914, samRNA-Spikebeta-TCE9
- GRT-R918, HIV-negative and PLWH, With and Without Prior Vaccination (Part D) (Experimental): Participants will be ≥18 and <60 years or ≥60 years, HIV-Negative and PLWH with no prior vaccination to SARS-CoV-2 (Cohorts D1, D2, D5, D6) or with prior vaccination to SARS-CoV-2 (Cohorts D3, D4, D7, D8). Cohorts will receive doses of GRT-R918 administered as prime and boost on Days 1 and 29, or as boost ≥2 months after prior SARS-CoV-2 vaccination. Parts B, C, and D will be run in parallel.
  Interventions: Drug: GRT-R918, samRNA-SpikeOmicron-N-TCE11

INTERVENTIONS:
Drug: GRT-R912, samRNA-Spikebeta-TCE11 — IM injection of GRT-R912. Doses will be decided after safety review of Part A.
  Arms: GRT-R912 or GRT-R914, People Living with HIV (PLWH) (Part C); GRT-R912, HIV-negative (Part B)
Drug: GRT-R914, samRNA-Spikebeta-TCE9 — Part A: 3 microgram (mcg), 10 mcg, or 30 mcg intramuscular (IM) injection of GRT-R914.
  Part C: IM injection of GRT-R914. Doses decided after safety review of Part A.
  Arms: GRT-R912 or GRT-R914, People Living with HIV (PLWH) (Part C); GRT-R914, HIV-negative (Part A)
Drug: GRT-R918, samRNA-SpikeOmicron-N-TCE11 — IM injection of GRT-R918. Doses will be decided after safety review of Part A.
  Arms: GRT-R918, HIV-negative and PLWH, With and Without Prior Vaccination (Part D)

SUMMARY:
The primary objective is to assess the safety and tolerability of samRNA vaccines GRT-R912, GRT-R914, and GRT-R918 when administered as prime and/or boost in healthy adult participants naïve to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), SARS-CoV-2 convalescent, previously vaccinated, or non-vaccinated participants, and people living with HIV (PLWH) or HIV-negative.

DETAILED DESCRIPTION:
This Phase 1 clinical trial (CORAL-CEPI) will assess the potential of second-generation Coronavirus Disease 2019 (COVID-19) vaccines. These vaccines use a codon optimized Spike (S) cassette with additional T cell epitopes (TCE) (cassette S-TCE) covering multiple epitopes from non-spike proteins to safely drive strong, broad, and durable B cell and T cell immune responses to SARS-CoV-2. This trial will assess the potential to generate B cell and T cell responses against SARS-CoV-2 in both people living with HIV (PLWH) and HIV-negative participants, in participants who have previously been infected by SARS-CoV-2, and those who are naive to SARS-CoV-2, meaning they have neither been infected with nor vaccinated against SARS-CoV-2. GRT-R912, GRT-R914, and GRT-R918 are vaccines using a samRNA vector based and administered as either a single dose or two dose regimen, providing an option for a potent, single-modality approach.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female at least 18 years and no more than 65 years of age at enrollment (Parts A, B, and C only).
* No previous SARS-CoV-2 infection or recovered.
* HIV-negative status confirmed by laboratory testing.

Additional inclusion criteria for PLWH:

* Serum positive HIV test or history of HIV infection.
* On anti-retroviral therapy for at least 3 months before screening and clinically stable.

Additional inclusion criteria for Part D (GRT-R918):

* Male or non-pregnant female between 18 and <60 years of age at enrollment.
* Male or non-pregnant female greater than or equal to 60 years of age at enrollment.
* Received any authorized SARS-CoV-2 vaccine series at least 2 months prior to study vaccine.

Exclusion Criteria:

* Current active infection with COVID-19.
* Positive for SARS-CoV-2 by nasal swab polymerase chain reaction (PCR) at screening.
* Currently receiving treatment or prevention agents with activity against SARS-CoV-2.
* Breastfeeding, pregnant, or planning to become pregnant during the course of the study.
* Received or plans to receive any non-study provided SARS-CoV-2 vaccine (including boost) during the study period (except for Part D).
* Received or plans to receive any live, attenuated vaccine within 28 days before or after study vaccination.
* Received or plans to receive any subunit or killed vaccine within 14 days before or after vaccination.
* Received or plans to receive immunoglobulins and/or any blood products within the 3 months preceding the planned administration of first study vaccination or at any time during the study.
* Currently active viral infection of hepatitis B virus or hepatitis C virus.

Additional exclusion criteria for PLWH:

* Screening CD4+ T cell count ≤200 cells/mcL.
* Viral load ≥10,000 virus particles/mL.
* History of opportunistic illness indicative of Stage 3 HIV infection.
* Acute febrile illness within 4 weeks before the first vaccination.

Additional exclusion criterion for Part D (GRT-R918) Cohorts D3, D4, D7, and D8:

- Received last dose of any authorized SARS-CoV-2 vaccine series within 2 months prior to study vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Solicited Local Reactogenicity Signs and Symptoms | Up to 7 days after vaccination
Number of Participants with One or More Solicited Systemic Reactogenicity Signs and Symptoms | Up to 7 days after vaccination
Number of Participants with Unsolicited Adverse Events | Up to 7 days after vaccination
Number of Participants with One or More Serious Adverse Events | Up to ~14 months after vaccination

SECONDARY OUTCOMES:
Response Rate of SARS-CoV-2 Specific Antibody Binding and Neutralization Titers in Serum Samples | Up to ~14 months after vaccination
Magnitude of SARS-CoV-2 Specific Antibody Binding and Neutralization Titers in Serum Samples | Up to ~14 months after vaccination
Response Rate of SARS-CoV-2 Specific CD4+ and CD8+ T cells by Intracellular Cytokine Staining (ICS) | Up to ~14 months after vaccination
Magnitude of SARS-CoV-2 Specific CD4+ and CD8+ T cell Response by ICS | Up to ~14 months after vaccination
Functional Profiling of SARS-CoV-2 Specific CD4+ and CD8+ T cells by ICS | Up to ~14 months after vaccination
Response Rate of SARS-CoV-2- Specific CD4+ and CD8+ T cells by Interferon-Gamma Enzyme-linked Immunospot (ELISpot) | Up to ~14 months after vaccination
Magnitude of SARS-CoV-2- Specific CD4+ and CD8+ T cell Response by Interferon-Gamma ELISpot | Up to ~14 months after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Martin, DO, Study Director — Gritstone bio, Inc.
Locations (4):
- South Africa (4):
  - Newtown Clinical Research Centre, Johannesburg
  - WITS RHI Shandukani Research Centre, Johannesburg
  - Wits Vaccines & Infections Diseases Analytics (VIDA) Research Unit, Johannesburg
  - Setshaba Research Center, Pretoria